CLINICAL TRIAL: NCT06676605
Title: Assessment of Ashwagandha Pills Consumption in the Amelioration of Obesity-associated Parameters in Mexican Adults with Overweight and Obesity
Brief Title: Impact of Ashwagandha in Obesity Parameters from Mexican Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ivan Luzardo-Ocampo (Other)
Collaborators: Tecnologico de Monterrey (Other); Universidad Autonoma de Nuevo Leon (Other)
Responsible Party: Sponsor-Investigator, Ivan Luzardo-Ocampo, Professor Researcher, Universidad Autonoma de Queretaro
Organization: Universidad Autonoma de Queretaro (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202301
Record Dates: First submitted 2024-11-01; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — Ashwagandha

STUDY DESIGN:
Intervention Model Description: This clinical trial was a double-blind, randomized, placebo-controlled study conducted in the Nutrition department with the Clinical Analysis Laboratory at University of Monterrey. It aimed to evaluate ashwagandha's effect on serum lipid concentrations and body composition in Mexican adults with overweight and obesity. Eligible participants were adults with a BMI of 25 kg/m^2 or higher, glucose levels around 100 mg/dL, LDL-C levels of 160 mg/dL or higher, total cholesterol levels of 200 mg/dL or higher, HDL-C levels lower than 40 mg/dL, and triglyceride levels exceeding 150 mg/dL. Participants provided informed consent per NOM-012-SSA3-2012 guidelines. They followed a prescribed dietary plan including 500 mg daily ashwagandha (Withania somnifera), authorized for use by the FDA. The supplementation period lasted 40 days. Participants were randomly assigned to the intervention group (W. somnifera, n=17) or placebo group (starch rice capsule/tablet, n=17).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: In this double-blind study, rigorous masking procedures were implemented to ensure the integrity of the results. None of the participants knew or met each other, and they had no prior information about the researcher conducting the study. Participants were instructed not to discuss their experiences, feelings, or outcomes with each other throughout the study duration. Furthermore, the researchers who processed the data were blinded to the participants' identities; they only analyzed the biochemical and anthropometric parameters without knowing which patient each set of data belonged to or any personal background information. This ensured that the analysis remained unbiased and confidential.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): The intervention group consisted of 17 participants who were administered a dietary supplement of Withania somnifera, classified as such and subject to FDA regulations comparable to pharmaceutical medications. Over a period of 40 days, participants in this group consumed 500 mg capsules of W. somnifera daily, in accordance with the manufacturer's instructions and within the recommended dose range of 240-600 mg. Prior to the supplementation period, comprehensive anthropometric and biochemical analyses were carried out to establish baseline measurements. Members of this group also received personalized meal plans to ensure that any observed changes were a direct result of the supplementation. Additionally, participants were closely monitored via email and/or text messages to remind them of study guidelines, address any questions or concerns, and watch for potential adverse effects.
  Interventions: Dietary Supplement: Withania somnifera
- Placebo Group (Placebo Comparator): The placebo group also comprised 17 participants who were given a capsule/tablet of starch rice daily for the same 40-day period. Like the intervention group, participants in the placebo group underwent initial anthropometric and biochemical analyses to set baseline measurements before starting the supplementation period. This group similarly received personalized meal plans to ensure that any observed changes could be accurately attributed to the placebo effect. The placebo group participants were monitored via email and/or text messages to reinforce study guidelines, answer any questions or concerns about their meal plans or supplements, and monitor for any potential adverse effects.
  Interventions: Other: Placebo Intervention

INTERVENTIONS:
Dietary Supplement: Withania somnifera — The experimental supplement administered to patients in this study was Withania somnifera, commonly known as ashwagandha. It is classified as a dietary supplement and is regulated similarly to pharmaceutical medications. The supplement has been authorized for commercialization and use by the Food and Drug Administration (FDA). Participants received the supplement in the form of 500 mg capsules, taken daily over a 40-day period, following the manufacturer's instructions. The range of the recommended daily dose is between 240 and 600 mg. The purpose of administering this supplement was to evaluate its impact on various health parameters, including serum lipid concentrations and body composition, in the study's participants.
  Other Names: Ashwagandha
  Arms: Intervention Group
Other: Placebo Intervention — The product administered to the placebo group was designed to simulate the appearance and administration of the experimental supplement but without containing any active ingredients. Participants in the placebo group received capsules/tablets filled with starch rice. These capsules were taken daily over the same 40-day period as the experimental group, ensuring that the placebo group followed identical administration and monitoring procedures. The use of starch rice capsules aimed to serve as a neutral control, allowing for a comparison between the effects of the actual Withania somnifera supplement and the placebo.
  Other Names: Pills
  Arms: Placebo Group

SUMMARY:
This clinical trial aimed to assess the impact of ashwagandha supplementation on serum lipid concentrations and body composition in Mexican adults with overweight and obesity. It was a double-blind, placebo-controlled pilot study, including adult patients who consumed ashwagandha pills for 40 days after giving informed consent. Two groups were part of the study: an experimental group receiving the supplement and a placebo group. Measurements conducted included anthropometric parameters and blood biochemical parameters.

DETAILED DESCRIPTION:
This clinical trial aimed to assess the impact of ashwagandha supplementation on serum lipid concentrations and body composition in Mexican adults with overweight and obesity through a double-blind, randomized, placebo-controlled protocol. The study included adult patients who met inclusion such as a Body Mass Index (BMI) of 25 kg/m^2 or higher, glucose levels around 100 mg/dL, LDL-C levels of 160 mg/dL or higher, total cholesterol levels of 200 mg/dL or higher, HDL-C levels lower than 40 mg/dL, and triglyceride levels exceeding 150 mg/dL). Patients were excluded if they were pregnant, had diabetes mellitus, hypertension, or hypersensitivity to Solanaceae products.

Volunteers signed an informed consent form as per NOM-012-SSA3-2012 guidelines, detailing the study's purpose and terms. Participants adhered to a prescribed dietary plan that included Ashwagandha (Withania somnifera) supplementation and consented to monitoring of their dietary intake and biochemical parameters measurement.

The ashwagandha supplementation involved 500 mg capsules taken daily for 40 days, with an intervention group (W. somnifera supplementation, 500 mg/day, n=17) and a placebo group (starch rice capsule/tablet/day, n=17). Both groups received personalized meal plans to ensure that observed changes were directly attributable to the supplements.

Anthropometric measurements included body weight, waist circumference, and BMI. Blood samples were extracted after 12 hours of fasting using a vacutainer system, and biochemical determinations were processed the same day with semi-automated equipment via COBAS® colorimetric methods. Parameters such as glucose, triglycerides, cholesterol, LDL-c, HDL-c, and VLDL-c were analyzed.

Sociodemographic data were described by gender, while clinical and anthropometric variables were categorized by intervention and control groups. Quantitative variables were compared using the student's t-test for related samples. Significant differences between baseline and experimental groups were found for total cholesterol, HDL, LDL, VLDL, the LDL/HDL-c ratio, and triglycerides.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who are willing to comply with the study guidelines for a 40-day period.
2. Individuals who consent to undergo initial anthropometric and biochemical analyses.
3. Participants willing to follow personalized meal plans.
4. Individuals who agree to receive reminders and monitoring communication via email and/or text messages.

Exclusion Criteria:

1. Individuals with known allergies or intolerances to Withania somnifera or starch rice.
2. Participants who are unable or unwilling to follow the daily supplementation regimen.
3. Individuals with medical conditions that might interfere with the study results or pose a health risk when taking the supplement.
4. Participants currently taking any other supplements or medications that could interfere with the study outcomes.

Ages: 29 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Body Weight Measurement | Along with the 40 days
  Measured body weight did not change between baseline and experimental groups.
Waist circumference | Along with the 40 days
  Measurement of waist circumference, that did not change statistically.
Diastolic blood pressure | Along with the 40 days
  Measurement of diastolic blood pressure, that did not change statistically.
Blood Glucose | Along with the 40 days
  Initial and final blood glucose only changed for the placebo group (p:0.008).
Blood lipids profile | Along with the 40 days
  Initial and final values of blood lipids profile parameters for each group changed statistically (Experimental: Total cholesterol, HDL-c, LDL-cm VLDL-c, LDL/HDL-c ratio, and triglycerides; Placebo: HDL-c, LDL-c, and LDL/HDL-c ratio)
Body Mass Index Measurement | Along with the 40 days]
  Quantified body mass index did not change between baseline and experimental groups

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Joanna Caballero-Prado, Ph. D., Principal Investigator — Universidad Autonoma de Nuevo Leon
Locations (1):
- Nutrition Department at Universidad Autonoma de Nuevo Leon, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No
Data will be shared after reasonable request and under permission by Bioethics Committee Board